CLINICAL TRIAL: NCT03508180
Title: Randomized Study Assessing the Benefits of Foot Reflexology in Patients With Gastrointestinal or Thoracic Cancer With Chemotherapy
Brief Title: Benefit Evaluation of Foot Reflexology in Oncology
Acronym: REFYO-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL17_0676
Record Dates: First submitted 2018-03-05; First posted 2018-04-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer and Cancer of Digestive System
Keywords: Supportive care; cancer; foot reflexology; nausea; vomiting
MeSH Terms: conditions — Lung Neoplasms; Digestive System Neoplasms; Neoplasms; Nausea; Vomiting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot reflexology (Experimental): patients WITH foot reflexology session during chemotherapy treatments
  Interventions: Behavioral: INTERVIONNAL
- platinum-based treatment (Placebo Comparator): Patients WITHOUT ANY foot reflexology session during chemotherapy treatments
  Interventions: Other: CONTROL

INTERVENTIONS:
Behavioral: INTERVIONNAL — Foot reflexology session (30 minutes) each course of chemotherapy (total 4 courses) during the 4 hours following the first 2 hours of injection + auto-massage done by the patient between each course.
  During a session focused on the treatment of nausea / vomiting, the reflexologist will stimulate the reflex zones related to the digestive system in order to calm and stimulate all areas for deep relaxation of the patient.
  Arms: foot reflexology
Other: CONTROL — None intervention.
  Arms: platinum-based treatment

SUMMARY:
Chemotherapy with platinum salts is very emetic. The aim of this study is to evaluate the benefits of foot reflexology in nausea and vomiting induced by platinum salts-based chemotherapy in patients with thoracic or digestive tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a thoracic or digestive cancer with indication of management with platinum salts-based chemotherapy
* Good performance status of (ECOG 0-2)
* More than 18 years old
* Ability to complete the questionnaires (comprehension oral and written French language) and to carry out the required exercises.
* Patient affiliated to Social Security or equivalent
* Informed consent signed

Exclusion Criteria:

* Phlebitis
* Cellar syndrome
* Weight loss> 5% in 3 months
* Uncontrolled pain
* Patients under morphine and derivatives
* Brain metastases
* Patient benefiting from foot reflexology outside the study
* Patient under guardianship or curatorship or deprived of his rights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of nausea and vomiting | 6 hours
  The relative change in VAS* associated with nausea and vomiting will be evaluated between T1 (measured at least 2 hours after the start of chemotherapy injection) and T2 (measured at least 6 hours after the start of injection of the drug chemotherapy).
  *VAS : from 0 to 10 ; 0 is no nausea or vomiting and 10 is insufferable nausea or vomiting

SECONDARY OUTCOMES:
Nausea and vomiting between each chemotherapy | Day 0, between day 14 and day 21, between day 28 and day 42, between day 42 and day 63.
  Between each chemotherapy the patient notes daily whether or not he has had nausea on a notebook.
Quality of life | Between day 0 and day 78
  Relative variation of the EORTC QLQC 30* (European Organisation for Research and Treatment of Cancer) between the inclusion visit (V2) and the end-of-study visit (V6).
  *EORTC QLQ C30 : All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Anxiety | Between day 0 and day 78
  Relative variation of the HADS* (Hospital and Anxiety Depression Scale) anxiety score between the inclusion visit (V2) and the end-of-study visit (V6).
  *HADS : 0 to 21, the highest scores corresponding to the presence of a more severe symptomatology
Body image | Day 0
  Evaluation of the body image to the end-of-study visit by the Body Image Questionnaire* (BIC), which measures the body image at a given moment t. The analysis will take into account the self-esteem assessed upon the inclusion visit on the Rosenberg scale** (V2).
  *BIC : The total score is between 19 and 95.
  **Rosenberg Scale : The total score ranges from 10 to 40. A score below 31 is considered low self-esteem

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Jean SOUQUET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France

REFERENCES:
- [Result] Murat-Ringot A, Souquet PJ, Chauvenet M, Rentler C, Subtil F, Schott AM, Preau M, Piriou V. The Effects of Foot Reflexology on Chemotherapy-Induced Nausea and Vomiting in Patients with Digestive System or Lung Cancer: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jul 14;9(7):e17232. doi: 10.2196/17232. PMID 32449505
- [Result] Murat-Ringot A, Souquet PJ, Subtil F, Boutitie F, Preau M, Piriou V. The Effect of Foot Reflexology on Chemotherapy-Induced Nausea and Vomiting in Patients With Digestive or Lung Cancer: Randomized Controlled Trial. JMIR Cancer. 2021 Nov 5;7(4):e25648. doi: 10.2196/25648. PMID 34738909